CLINICAL TRIAL: NCT03920293
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of Ravulizumab in Complement-Inhibitor-Naïve Adult Patients With Generalized Myasthenia Gravis
Brief Title: Safety and Efficacy Study of Ravulizumab in Adults With Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALXN1210-MG-306; 2018-003243-39 (EudraCT Number)
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Results first posted 2022-05-26 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-04

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: All investigative site personnel, sponsor staff, sponsor designees, staff directly associated with the conduct of the study, and all participants will be blinded to treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ravulizumab (Experimental): Participants will receive ravulizumab for the duration of the study.
  Interventions: Biological: Ravulizumab
- Placebo (Placebo Comparator): Participants will receive placebo during the 26-week randomized-controlled period of the study, after which they will enter the open-label extension period of the study and receive ravulizumab.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ravulizumab — Concentrated sterile, preservative-free aqueous solution (10 milligrams [mg]/milliliter [mL]) in single-use, 30-mL vial for intravenous (IV) infusion. Single loading dose on Day 1, followed by regular maintenance dosing beginning on Day 15, based on weight.
  Other Names: ALXN1210; Ultomiris
  Arms: Ravulizumab
Drug: Placebo — Matching, sterile, preservative-free aqueous solution in single-use, 30-mL vial for IV infusion. Single loading dose on Day 1, followed by regular maintenance dosing beginning on Day 15, based on weight.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of ravulizumab for the treatment of participants with generalized myasthenia gravis (gMG).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Myasthenia Gravis at least 6 months (180 days) prior to the date of the Screening Visit as confirmed by specific criteria.
2. Myasthenia Gravis Foundation of America Clinical Classification Class II to IV at screening.
3. MG-ADL profile must be ≥ 6 at screening and randomization (Day 1).
4. Vaccinated against meningococcal infections within 3 years prior to, or at the time of, initiating study drug to reduce the risk of meningococcal infection (N meningitidis).

Exclusion Criteria:

Medical Conditions

1. Any active or untreated thymoma. History of thymic carcinoma or thymic malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥ 5 years before screening.
2. History of thymectomy within the 12 months prior to screening.
3. History of N meningitidis infection.
4. Use of the following within the time period specified below:

   * IV immunoglobulin within 4 weeks of randomization
   * Use of plasma exchange within 4 weeks of randomization
   * Use of rituximab within 6 months of screening
5. Participants who have received previous treatment with complement inhibitors (for example, eculizumab).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (99):
- United States (46):
  - Research Site, Phoenix, Arizona
  - Research Site, Irvine, California
  - Research Site, Loma Linda, California
  - Research Site, Palo Alto, California
  - Research Site, San Francisco, California
  - Research Site, Sylmar, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Fairfield, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Rolling Meadows, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Burlington, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, East Lansing, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Columbia, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Great Neck, New York
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Richmond, Virginia
  - Research Site, Morgantown, West Virginia
- Research Site, Vienna, Austria
- Canada (4):
  - Research Site, Edmonton, Alberta
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (3):
  - Research Site, Brno
  - Research Site, Ostrava
  - Research Site, Prague
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Arhus C
  - Research Site, Copenhagen
- France (4):
  - Research Site, Garches
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Nice
- Germany (6):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Münster
  - Research Site, Würzburg
- Israel (2):
  - Research Site, Haifa
  - Research Site, Tel Aviv
- Italy (6):
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Rome
- Japan (13):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Hanamaki-shi
  - Research Site, Kawagoe-shi
  - Research Site, Moriguchi-shi
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Ube-shi
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Leiden
- Research Site, Porto, Portugal
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Seoul
  - Research Site, Yangsan
- Spain (4):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Murcia
- Research Site, Zurich, Switzerland

REFERENCES:
- [Derived] Vu T, Meisel A, Mantegazza R, Annane D, Katsuno M, Aguzzi R, Enayetallah A, Beasley KN, Rampal N, Howard JF. Terminal Complement Inhibitor Ravulizumab in Generalized Myasthenia Gravis. NEJM Evid. 2022 May;1(5):EVIDoa2100066. doi: 10.1056/EVIDoa2100066. Epub 2022 Apr 26. PMID 38319212
- [Derived] Meisel A, Annane D, Vu T, Mantegazza R, Katsuno M, Aguzzi R, Frick G, Gault L, Howard JF Jr; CHAMPION MG Study Group. Long-term efficacy and safety of ravulizumab in adults with anti-acetylcholine receptor antibody-positive generalized myasthenia gravis: results from the phase 3 CHAMPION MG open-label extension. J Neurol. 2023 Aug;270(8):3862-3875. doi: 10.1007/s00415-023-11699-x. Epub 2023 Apr 27. PMID 37103755
- [Derived] Vu T, Ortiz S, Katsuno M, Annane D, Mantegazza R, Beasley KN, Aguzzi R, Howard JF Jr. Ravulizumab pharmacokinetics and pharmacodynamics in patients with generalized myasthenia gravis. J Neurol. 2023 Jun;270(6):3129-3137. doi: 10.1007/s00415-023-11617-1. Epub 2023 Mar 9. PMID 36890354
- [Derived] Vanoli F, Mantegazza R. Ravulizumab for the treatment of myasthenia gravis. Expert Opin Biol Ther. 2023 Mar;23(3):235-241. doi: 10.1080/14712598.2023.2185131. Epub 2023 Mar 8. PMID 36852670
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1210-MG-306&attachmentIdentifier=f164e5fa-8534-413e-a765-e3c6b87e017c&fileName=ALXN1210-MG-306_CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized 1:1 to either the ravulizumab or placebo group during the Randomized-Controlled Period. Following the placebo-controlled part of the study, participants were transitioned to the ongoing Open-Label Extension Period to receive treatment with ravulizumab.
Groups:
- Ravulizumab to Ravulizumab: Participants received a weight-based single loading dose (2400 to 3000 mg) of ravulizumab IV on Day 1, followed by regular maintenance IV weight-based doses (3000 to 3600 mg) of ravulizumab beginning on Day 15 q8w during the 26-week Randomized-Controlled Period of the study. After the randomized-controlled part of the study, participants were transitioned to the ongoing open-label extension period to receive treatment with ravulizumab IV for up to 2 years.
- Placebo to Ravulizumab: Participants received a weight-based single loading dose of placebo IV on Day 1, followed by regular maintenance IV weight-based doses of placebo beginning on Day 15 q8w, during the 26-week Randomized-Controlled Period of the study. After the randomized-controlled part of the study, participants were transitioned to the ongoing open-label extension period to receive treatment with ravulizumab IV for up to 2 years.
Period: Randomized-Controlled Period
Arm/Group | Ravulizumab to Ravulizumab | Placebo to Ravulizumab
Started | 86 | 89
Received at Least 1 Dose of Study Drug | 86 | 89
Completed | 79 | 83
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Sponsor Decision | 0 | 1
Not completed — Death | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Noncompliance | 1 | 0
Period: Open- Label Extension Period
Arm/Group | Ravulizumab to Ravulizumab | Placebo to Ravulizumab
Started | 78 | 83
Completed | 60 | 63
Not Completed | 18 | 20
Not completed — Participants who transitioned to alternative treatment by the Investigator when the study closed | 3 | 5
Not completed — Death | 3 | 3
Not completed — Physician Decision | 5 | 3
Not completed — Withdrawal by Subject | 7 | 9

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All randomized participants who received at least 1 dose of study drug.
Groups:
- Ravulizumab: Participants received a weight-based single loading dose (2400 to 3000 mg) of ravulizumab IV on Day 1, followed by regular maintenance IV weight-based doses (3000 to 3600 mg) of ravulizumab beginning on Day 15 q8w during the 26-week Randomized-Controlled Period of the study. After the randomized-controlled part of the study, participants were transitioned to the ongoing open-label extension period to receive treatment with ravulizumab IV for up to 2 years.
- Placebo: Participants received a weight-based single loading dose of placebo IV on Day 1, followed by regular maintenance IV weight-based doses of placebo beginning on Day 15 q8w, during the 26-week Randomized-Controlled Period of the study. After the randomized-controlled part of the study, participants were transitioned to the ongoing open-label extension period to receive treatment with ravulizumab IV for up to 2 years.
- Total: Total of all reporting groups
Arm/Group | Ravulizumab | Placebo | Total
Number analyzed (Participants) | 86 | 89 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (13.82) | 53.3 (16.05) | 55.6 (15.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 45 | 89
  Male | 42 | 44 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 79 | 78 | 157
  Unknown or Not Reported | 5 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 15 | 16 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 67 | 61 | 128
  Other | 0 | 1 | 1
  Unknown or Not Reported | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Myasthenia Gravis-Activities Of Daily Living (MG-ADL) Total Score At Week 26
Description: The MG-ADL is an 8-point questionnaire that focused on relevant symptoms and functional performance of activities of daily living in participants with MG. The 8 items of the MGADL questionnaire were derived from symptom-based components of the original 13-item QMG scale to assess disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects from MG. In this functional status instrument, each response was graded 0 (normal) to 3 (most severe). The range of total MG-ADL score was 0 to 24. A decrease in score indicated improvement. Estimates were based on Mixed Effect Repeated Measures (MMRM) that included treatment group, stratification factor region, and MG-ADL total score at baseline, study visit, and study visit by treatment group interaction.
Time Frame: Baseline, Week 26
Population: Full Analysis Set: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 86 | 89
units on a scale | -3.1 (0.38) | -1.4 (0.37)
Statistical Analysis 1: Comparison: Ravulizumab vs Placebo; Test type: Superiority; p = 0.0009, MMRM — Statistical significance was tested at α=0.05; LS Mean Difference = -1.6, 95% CI 2-sided [-2.6 to -0.7], Standard Error of Mean 0.49

2. Secondary Outcome: Change From Baseline In The Quantitative Myasthenia Gravis (QMG) Total Score At Week 26
Description: The QMG scoring system consisted of 13 items: ocular (2 items), facial (1 item), bulbar (2 items), gross motor (6 items), axial (1 item), and respiratory (1 item); each graded 0 to 3, with 3 being the most severe. The range of total QMG score is 0 to 39. The QMG scoring system was considered to be an objective evaluation of therapy for MG and was based on quantitative testing of sentinel muscle groups. A decrease in score indicated improvement. Estimates were based on MMRM that included treatment group, stratification factor region, and QMG total score at baseline, study visit, and study visit by treatment group interaction.
Time Frame: Baseline, Week 26
Population: Full Analysis Set: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 86 | 89
units on a scale | -2.8 (0.46) | -0.8 (0.45)

3. Secondary Outcome: Percentage of Participants With a Quantitative Myasthenia Gravis (QMG) Total Score Reduction of at Least 5 Points At Week 26
Description: The QMG scoring system consisted of 13 items: ocular (2 items), facial (1 item), bulbar (2 items), gross motor (6 items), axial (1 item), and respiratory (1 item); each graded 0 to 3, with 3 being the most severe. The range of total QMG score is 0 to 39. A decrease in score indicated improvement. Percentage of participants with a ≥5-point reduction in the QMG total score are reported. Estimates were based on a generalized linear mixed model (GLMM) that included treatment group, stratification factor region and QMG total score at baseline, study visit and study visit by treatment group interaction.
Time Frame: Week 26
Population: Full Analysis Set: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 86 | 89
percentage of participants | 30.0 [19.2 to 43.5] | 11.3 [5.6 to 21.5]

4. Secondary Outcome: Change From Baseline In the Revised 15 Component Myasthenia Gravis Quality of Life (MG-QOL15r) At Week 26
Description: The revised Myasthenia Gravis Qualify of Life 15-item scale (MG-QOL15r) is a health-related QoL evaluative instrument specific to participants with MG. The MG-QOL15r was designed to provide information about participants' perception of impairment and disability, determine the degree to which disease manifestations are tolerated, and to be administered and interpreted easily. Each item was graded on a scale of 0 to 2, with 2 being the most severe. The range of MG-QOL15r score is 0 to 30. Higher scores indicated greater extent of and dissatisfaction with MG-related dysfunction. Estimates are based on MMRM that included treatment group, stratification factor region and MG-QOL15r score at baseline, study visit and study visit by treatment group interaction.
Time Frame: Baseline, Week 26
Population: Full Analysis Set: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 86 | 89
score on a scale | -3.3 (0.71) | -1.6 (0.70)

5. Secondary Outcome: Change From Baseline in Neurological Quality of Life (Neuro-QoL) Fatigue Score at Week 26
Description: The Neuro-QOL Fatigue is a reliable and validated brief 19-item survey of fatigue, completed by the participant. Each items was rated on a scale of 1 to 5, with 5 being the most severe. The range of total score is 19 to 95. Higher scores indicated greater fatigue and greater impact of MG on activities. Estimates were based on MMRM that included treatment group, stratification factor region and Neuro-QoL Fatigue score at baseline, study visit, and study visit by treatment group interaction.
Time Frame: Baseline, Week 26
Population: Full Analysis Set: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 86 | 89
units on a scale | -7.0 (1.92) | -4.8 (1.87)

6. Secondary Outcome: Percentage of Participants With a Myasthenia Gravis Activities of Daily Living (MG-ADL) Total Score Reduction of at Least 3 Points At Week 26
Description: The MG-ADL is an 8-point questionnaire that focused on relevant symptoms and functional performance of activities of daily living in participants with MG. The 8 items of the MGADL questionnaire were derived from symptom-based components of the original 13-item QMG scale to assess disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects from MG. In this functional status instrument, each response was graded 0 (normal) to 3 (most severe). The range of total MG-ADL score was 0 to 24. A decrease in score indicated improvement. Percentage of participants with a ≥3-point reduction in the MG-ADL total score are reported. Estimates were based on a GLMM that included treatment group, stratification factor region and MG-ADL total score at baseline, study visit and study visit by treatment group interaction.
Time Frame: Week 26
Population: Full Analysis Set: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab | Placebo
Number analyzed (Participants) | 86 | 89
percentage of participants | 56.7 [44.3 to 68.3] | 34.1 [23.8 to 46.1]

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) up to 2 years
Description: Treatment-emergent adverse events were reported for 26-week randomized-controlled period and open-label extension period separately.
Groups:
- Randomized-Controlled Period: Ravulizumab: Participants received a weight-based single loading dose (2400 to 3000 mg) of ravulizumab IV on Day 1, followed by regular maintenance IV weight-based doses (3000 to 3600 mg) of ravulizumab beginning on Day 15 q8w during the 26-week Randomized-Controlled Period of the study.
- Randomized-Controlled Period: Placebo: Participants received a weight-based single loading dose of placebo IV on Day 1, followed by regular maintenance IV weight-based doses of placebo beginning on Day 15 q8w, during the 26-week Randomized-Controlled Period of the study.
- Open-Label Extension Period: Placebo to Ravulizumab: After the randomized-controlled part of the study, participants in the placebo group were transitioned to the ongoing open-label extension period to receive treatment with ravulizumab IV for up to 2 years.
- Open-Label Extension Period: Ravulizumab to Ravulizumab: After the randomized-controlled part of the study, participants in the ravulizumab group were transitioned to the ongoing open-label extension period to receive treatment with ravulizumab IV for up to 2 years.
Arm/Group | Randomized-Controlled Period: Ravulizumab | Randomized-Controlled Period: Placebo | Open-Label Extension Period: Placebo to Ravulizumab | Open-Label Extension Period: Ravulizumab to Ravulizumab
All-Cause Mortality (participants affected / at risk) | 2/86 | 0/89 | 3/83 | 3/78
Serious Adverse Events (participants affected / at risk) | 20/86 | 14/89 | 32/83 | 24/78
Other Adverse Events (participants affected / at risk) | 77/86 | 75/89 | 79/83 | 77/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized-Controlled Period: Ravulizumab (N=86) | Randomized-Controlled Period: Placebo (N=89) | Open-Label Extension Period: Placebo to Ravulizumab (N=83) | Open-Label Extension Period: Ravulizumab to Ravulizumab (N=78)
COVID-19 pneumonia (Infections and infestations) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (4) | 4 (6)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis crisis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 3 (3) | 1 (2) | 4 (4)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion-related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Steroid diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gonococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neisseria infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic cystadenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vein rupture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized-Controlled Period: Ravulizumab (N=86) | Randomized-Controlled Period: Placebo (N=89) | Open-Label Extension Period: Placebo to Ravulizumab (N=83) | Open-Label Extension Period: Ravulizumab to Ravulizumab (N=78)
COVID-19 (Infections and infestations) | 5 (5) | 3 (3) | 26 (28) | 30 (32)
Urinary tract infection (Infections and infestations) | 5 (7) | 4 (5) | 8 (13) | 7 (9)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (7) | 11 (18) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 11 (15) | 10 (12) | 6 (6)
Nausea (Gastrointestinal disorders) | 9 (12) | 9 (10) | 9 (18) | 7 (8)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 0 (0) | 4 (5) | 4 (4)
Headache (Nervous system disorders) | 16 (19) | 23 (27) | 17 (21) | 12 (19)
Dizziness (Nervous system disorders) | 8 (9) | 3 (3) | 6 (10) | 4 (5)
Fatigue (General disorders) | 6 (7) | 6 (6) | 6 (7) | 7 (7)
Pyrexia (General disorders) | 1 (1) | 5 (6) | 5 (5) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5) | 10 (10) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 7 (8) | 9 (15) | 11 (14)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 9 (9) | 2 (4)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (6)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 5 (6) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 10 (11) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (6) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (7)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 7 (8) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 5 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT03920293/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT03920293/SAP_001.pdf